CLINICAL TRIAL: NCT05525884
Title: Mechanism of Serum PRL in the Development of MAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shen Qu (Other)
Responsible Party: Sponsor-Investigator, Shen Qu, Principle investigator, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: PRL
Record Dates: First submitted 2021-12-15; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Type2 Diabetes; Fatty Liver, Nonalcoholic; Liver Fibrosis
Keywords: Type 2 Diabetes; Metabolic associated fatty liver disease,; Prolactin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MAFLD and Non-MAFLD
  Interventions: Other: non-invasive method, Fibroscan
- Steatosis and Non-Steatosis
  Interventions: Other: non-invasive method, Fibroscan
- Fibrosis and Non-Fibrosis
  Interventions: Other: non-invasive method, Fibroscan

INTERVENTIONS:
Other: non-invasive method, Fibroscan — Liver Ultrasound and transient elastography (FibroScan®)

SUMMARY:
Metabolic associated fatty liver disease (MAFLD) has currently reached a worldwide epidemic. Serum PRL levels within or outside physiological range have been found to affect metabolic homeostasis differently. However, the relationship between serum PRL and MAFLD among diabetic patients is unclear. The investigators aimed to explore the association between serum PRL and the risk of MAFLD in patients with type 2 diabetes (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* aged 18~65 years old,
* underwent the laboratory tests, hepatic ultrasonography, and valid transient elastography (FibroScan) examination

Exclusion Criteria:

* other known chronic liver diseases, such as chronic hepatitis B or C, autoimmune hepatitis, and haemochromatosis
* pre-existing active cancer, renal dysfunction, severe liver dysfunction, congestive heart failure or free abdominal fluid
* history of hyperthyroidism or hypothyroidism, pituitary diseases, and other types of diabetes
* significant alcohol consumption
* pregnancy
* receiving any therapeutic methods that could lead to liver steatosis or fibrosis, influence the glucolipid metabolism, or PRL levels, such as lipid-lowering, and PRL-lowering agents (bromocriptine) within 6 months prior to this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM who met the inclusion and criteria criteria were consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of MAFLD proposed by the international expert consensus statement in 2020 | 2019-2024
  MAFLD was diagnosed based on evidence of ultrasonically diagnosed hepatic steatosis in addition to one of the three criteria proposed by the international expert consensus statement in 2020, namely overweight/obesity, T2DM, or metabolic dysregulation regardless of alcohol consumption or other concomitant liver diseases. Metabolic dysregulation was defined by the presence of at least two metabolic risk abnormalities found in lean or normal weight patients, including hypertension, dyslipidemia, hyperglycemia, IR, and high CRP levels.
PRL | 2019-2024
  serum prolactin levels
High PRL (HP) | 2019-2024
  HP was defined as serum PRL ≥ 324mIU/L in males or ≥ 496mIU/L in females according to the normal reference value of serum PRL in our hospital.
Normal PRL (NP) | 2019-2024
  NP was defined as serum PRL < 324mIU/L in males or < 496mIU/L in females.
Diagnosis of hepatic steatosis | 2019-2024
  Those who have hepatic steatosis if CAP value ≥ 248 dB/m, which was obtained from transient elastography (FibroScan®) using the M probe or the XL probe.
Diagnosis of significant hepatic fibrosis | 2019-2024
  those who have significant hepatic fibrosis if LSM ≥ 7.0 kPa and ≥ 6.2 kPa (using either M or XL probes)

SECONDARY OUTCOMES:
Homeostasis model assessment of IR (HOMA-IR) | 2019-2024
  HOMA-IR was calculated as described by Matthews et al: FPG (mmol/L) × FINS (mU/L) /22.5.
Hypertension | 2019-2024
  it was defined by blood pressure ≥130/85mmHg or antihypertensive drugs.
Dyslipidemia | 2019-2024
  it was defined by plasma TG ≥ 1.7mmol/L in the total population or plasma HDL-C < 1.0 mmol/L for men and < 1.3 mmol/L for women, or specific drug treatment.
Overweight or obesity | 2019-2024
  it was defined as BMI ≥ 23 kg/m2 in Asians.
Abdominal obesity | 2019-2024
  It was diagnosed when WC ≥ 90/80 cm in Asian men and women.
T2DM | 2019-2024
  it was diagnosed according to the guideline for the prevention and treatment of T2DM in China (2020 edition)
High CRP | 2019-2024
  plasma CRP > 2 mg/L
High HOMA-IR | 2019-2024
  HOMA-IR≥ 2.5

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China